CLINICAL TRIAL: NCT04106687
Title: A Randomized Controlled Trial of Sacral Erector Spinae Block Versus Caudal Block for Postoperative Analgesia After Hypospadias Surgery in Children
Brief Title: Comparison Sacral Erector Spinae Block Versus Caudal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: Kocaeli University (Other); Koç University (Other)
Responsible Party: Principal Investigator, Gözen Öksüz, Assistant Professor, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019/12-16
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: All Children will be randomly assigned to one of 2 groups of 20 patients each using a computer-generated number table.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal Block (Active Comparator): After preoxygenation for three minutes, anesthesia would be induced with 8% sevoflurane inhalation in 50% oxygen and % 50 air ; 1ug/kg fentanyl and 3 mg/kg propofol is administered intravenously. Then laryngeal mask is inserted when conditions are satisfactory ultrasound guided caudal block wil performe with bupivacaine 1 ml/kg as 0.25%.
  Interventions: Procedure: Ultrasound Guided Caudal Block; Procedure: Sacral Erector Spinae Block
- Sacral Erector Spinae Block (Active Comparator): After preoxygenation for three minutes, anesthesia would be induced with 8% sevoflurane inhalation in 50% oxygen and % 50 air ; 1ug/kg fentanyl and 3 mg/kg propofol is administered intravenously. Then laryngeal mask is inserted when conditions are satisfactory ultrasound guided sacral erector spinae block wil performe with bupivacaine 1 ml/kg as 0.25%.
  Interventions: Procedure: Ultrasound Guided Caudal Block; Procedure: Sacral Erector Spinae Block

INTERVENTIONS:
Procedure: Ultrasound Guided Caudal Block — Postoperative pain procedure
Procedure: Sacral Erector Spinae Block — Postoperative pain procedure

SUMMARY:
The purpose of this research study is to find the best way to decrease pain in children whom have had hypospadias surgery. Investigators will perform two technique; Caudal block or Sacral erector spinae block.

The results of this study will help learn how to best control pain in children having surgery hypospadias surgery.

DETAILED DESCRIPTION:
Children aged 1-9 years undergoing hypospadias surgeries would be recruited in this randomized study.

Children would be monitored by electrocardiogram, pulse oximeter and non-invasive blood pressure.

After preoxygenation for three minutes, anesthesia would be induced with 8% sevoflurane inhalation in 50% oxygen and % 50 air ; 1ug/kg fentanyl and 3 mg/kg propofol is administered intravenously. Then laryngeal mask is inserted when conditions are satisfactory (jaw relaxed, lash reflex disappeared, no coughing, gagging, swallowing).After ethical committee approval, informed written consent will be obtained from all patients.

Consenting patients scheduled to have hypospadias surgery will be randomised to sacral erector spinae block or caudal block at the begin of surgery.

All patients heart rate,MAP and Oxygen saturation record intraoperatively. All patients will receive paracetamol if requirement for postoperative analgesia.All patient will transfer from PACU to day-surgery unit (DSU) if they achieved Modified Aldrete Score of ten.

All patients will be assessed postoperatively by a blinded investigator: in the postanesthesia care unit and at 30 min 1,2, 4, 6, 12, 24, hour postoperatively.FLACC score will be used.

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-9
2. ASA physical status I-II
3. Undergoing unilateral low abdominal surgery

Exclusion Criteria:

1. History of developmental delay or mental retardation, which will make observational pain intensity assessment difficult
2. Parent refusal
3. History of allergic reactions to local anesthetics
4. Rash or infection at the injection site
5. Anatomical abnormality
6. Bleeding diatheses
7. Coagulopathy
8. History of diseases renal hepatic cardiac upper or lower airway neurologica

Ages: 1 Year to 9 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2019-09-27 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Number of analgesic consumption | 24 hour
  Acetaminophen and Fentanly

SECONDARY OUTCOMES:
Face, Legs, Activity, Cry and Consolability Score (FLACC) | 24 hour
  FLACC scale will be used. The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain. The scale has five criteria, which are each assigned a score of 0, 1 or 2. FLACC scale will be recorded at postoperative 30 minute, 1,2,4,6,12,24 hour
Parent satisfaction scores | 24 hour
  By investigators until hospital discharge, then through telephone interview with parents after that. Will be scored between 1-3 (1- very bad, 2-good, 3-very good).

CONTACTS AND LOCATIONS:
Overall Officials: Can Aksu, M.D., Principal Investigator — Kocaeli University; Yavuz Gürkan, Professor, Principal Investigator — Koç University
Locations (3):
- Turkey (Türkiye) (3):
  - Koç University Hospital, Istanbul
  - Kahramanmaras Sutcu Imam University Hospital, Kahramanmaraş
  - Kocaeli University Hospital, Kocaeli

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oksuz G, Arslan M, Bilal B, Gisi G, Yavuz C. Ultrasound guided sacral erector spinae block for postoperative analgesia in pediatric anoplasty surgeries. J Clin Anesth. 2020 Mar;60:88. doi: 10.1016/j.jclinane.2019.08.006. Epub 2019 Sep 3. No abstract available. PMID 31491727
- [Background] Aksu C, Gurkan Y. Sacral Erector Spinae Plane Block with longitudinal midline approach: Could it be the new era for pediatric postoperative analgesia? J Clin Anesth. 2020 Feb;59:38-39. doi: 10.1016/j.jclinane.2019.06.007. Epub 2019 Jun 13. No abstract available. PMID 31203111